CLINICAL TRIAL: NCT07382297
Title: Analgesic Efficacy of Adding Ultra Sound Guided IPACK Block to Adductor Canal Block for Postoperative Pain Management After Excision of Tumors Around Knee: a Randomized Controlled Trial
Brief Title: Effect of Adding Ultrasound Guided IPACK Block to Adductor Canal Block for Postoperative Pain in Knee Tumor Excision
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AP2407-201-011
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-08

CONDITIONS: Cancer Pain
MeSH Terms: conditions — Cancer Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- adductor canal block with iPACK (Active Comparator): The adductor canal will be identified. a spinal needle 22 gauge x 3.5 inches will be advanced with the guidance of ultrasound in an in-plane technique, and 15ml of 0.5% bupivacaine will be injected then IPACK block will be performed The probe will be applied to the popliteal fossa for identification of the popliteal artery and femur. Then, the probe will be slid distally for revealing the two femoral condyles followed by proximal sliding of the probe until the humps of the femoral condyles disappeared and the flat metaphysis appeared. a spinal needle 22G x 3.5 inches will be advanced from the lateral aspect and directed across the space between the popliteal artery and femur and once the needle reaches the medial edge of the femur, nearly at the level of the popliteal artery, negative aspiration will be confirmed and 15ml of 0.5% bupivacaine will be injected incrementally as the needle will be withdrawn.
  Interventions: Procedure: adductor canal block with iPACK
- control group (Other): visualizing the adductor canal without doing any block for the control group
  Interventions: Other: control group

INTERVENTIONS:
Procedure: adductor canal block with iPACK — The adductor canal will be identified. a spinal needle 22 gauge x 3.5 inches will be advanced with the guidance of ultrasound in an in-plane technique ,and 15ml of 0.5% bupivacaine will be injected then IPACK block will be performed. The probe will be applied to the popliteal fossa for identification of the popliteal artery and femur. Then, the probe will be slid distally for revealing the two femoral condyles followed by proximal sliding of the probe until the humps of the femoral condyles disappeared and the flat metaphysis appeared. a spinal needle 22G x 3.5 inches will be advanced from the lateral aspect and directed across the space between the popliteal artery and femur and once the needle reaches the medial edge of the femur, nearly at the level of the popliteal artery, negative aspiration will be confirmed and 15ml of 0.5% bupivacaine will be injected incrementally as the needle will be withdrawn
  Arms: adductor canal block with iPACK
Other: control group — The probe will be positioned at the midpoint between the anterior superior iliac spine and the upper pole of the patella.
  The adductor canal, which is a hyperechoic structure situated beneath the sartorius muscle, will be identified but no block will be done
  Arms: control group

SUMMARY:
the aim of this study is to determine the analgesic effect of iPACK in combination to ACB after the excision of tumors around the Knee regarding the following:

* Time to the 1st rescue analgesia.
* Postoperative morphine consumption.
* Postoperative visual analogue scale (VAS). This study will include patients, aged 18 to 65 years, belonging to the American Society of Anesthesiologists (ASA) physical status II to IV , undergoing excision of tumors around the knee under spinal anesthesia.

Patients will be randomly allocated Group iPACK plus Adductor canal block (ACB) : patients will receive ACB plus iPACK block.

• Control group : patients will not receive any block but will take morphine 3mg bolus at VAS more than 4 and regular NSAIDS and paracetamol iv.

DETAILED DESCRIPTION:
Immediate alleviation of postoperative pain after knee surgeries is critical for patients' postoperative recovery. Ineffective pain management may result in an extended hospital stay and rehabilitation period, as well as the development of chronic pain Non-opioid analgesics are insufficient to alleviate the pain that is intended to be relieved.

Although using Opioids have concerns regarding their potential side effects, which encompass nausea, vomiting, respiratory depression, and addiction Multimodal analgesia, which may include preemptive analgesia, neuraxial blockade, peripheral nerve block, and narcotic and non-narcotic analgesics, is an optimal approach for the management of acute pain following knee surgeries Adductor canal block (ACB) is an interfascial plane infiltration of local anesthetic used to block a portion of the saphenous nerve, which originates in the adductor canal, as well as the obturator nerve ACB combined with an iPACK block results in significantly better postoperative visual analog scale (VAS) scores, knee ranges of motion, as well as ambulation distances compared with ACB alone

ELIGIBILITY:
Inclusion Criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study
* American Society of Anesthesiologists (ASA) physical status II-IV.
* Patients undergoing excision of tumors around the knee under spinal anesthesia

Exclusion Criteria:

* Patient refusal.
* Neuromuscular disorders
* Allergy to local anesthetics
* Previous history of knee surgery
* Patients with a prior knee infection
* Contraindications to spinal anesthesia as coagulopathies and severe aortic stenosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Time to the 1st rescue analgesia | 24 hours postoperative
  Time to the 1st rescue analgesia

SECONDARY OUTCOMES:
Total morphine consumption | first 24 hour
  morphine consumed in 1st 24 hours postoperative in mg
pain score ( visual analogue scale) | at 2 hours ,4 hours,6 hours, 12 hours,18 hours and 24 h postoperatively
  assessment of postoperative pain using the visual analogue scale score. the scale is a straight horizontal line (100 mm). The ends are defined as the extreme limits of pain orientated from the left (no pain) to the right (worst pain).The patient marks on the line the point that they feel represents their perception of their current state.
  The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks.higher VAS score means worse pain

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Gamal Eldin Elsayed, MD, Study Director — National Cancer Institute (NCI)
Locations (1):
- National cancer institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No